CLINICAL TRIAL: NCT04177628
Title: Shared Decision Making With Breast Cancer Patients Offered Adjuvant Radiotherapy
Brief Title: Shared Decision Making With Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Danish Breast Cancer Cooperative Group (Other); University of Southern Denmark (Other); Danish Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DBCG RT SDM
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Shared Decision Making; Breast Neoplasms; Radiotherapy, Adjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Half the doctors at each center will receive training in SDM. These doctors will practice SDM supported by the in-consultation PtDA during every consultation in this study. The other half of the doctors will continue usual practice of informing the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Shared decision making (Experimental): Patients will be informed by a doctor randomized to practice shared decision making and use the in-consultation PtDA during the consultation on adjuvant radiotherapy.
  Interventions: Behavioral: Shared decision making supported by an in-consultation patient decision aid
- Arm B: Usual practice (No Intervention): Patients will be informed by a doctor randomized to inform about adjuvant radiotherapy according to usual practice.

INTERVENTIONS:
Behavioral: Shared decision making supported by an in-consultation patient decision aid — After having received training in SDM, the doctor will practice SDM supported by an in-consultation PtDA during the consultation with the participant.
  Arms: Arm A: Shared decision making

SUMMARY:
The aim of this project is to elucidate whether the use of shared decision making will influence patient engagement in the decision making process about adjuvant radiotherapy after breast conserving surgery for local breast cancer or early stages of local breast cancer.

DETAILED DESCRIPTION:
The risk of recurrence of breast cancer is lowered by adjuvant medical treatment as well as by radiotherapy (RT). On the other hand, all adjuvant treatments involve a risk of side effects; some are acute and transient while others are long-term. Considering the well-known side effects of irradiation, it seems appropriate to involve patients in the decision on whether to receive irradiation.

In the shared decision making (SDM) process clinicians and patients work together to make appropriate health decisions based on clinical evidence and the patient's informed preferences. A patient decision aid (PtDA) is instrumental in the SDM process.

This study is a multicenter, national trial randomizing doctors to either use or not use SDM and a PtDA when informing the patients about benefits and risks of receiving adjuvant radiotherapy.

It is not expected that significantly less patients will receive radiotherapy as a consequence of SDM. The primary aim of the study is to evaluate whether patient engagement in decision making is affected by SDM and the use of an in-consultation PtDA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified breast cancer or ductal carcinoma in situ breast cancer
* Candidate for adjuvant radiotherapy Danish Breast Cancer Group type F after breast-conserving surgery for T1-2, N0-Nmi, M0 disease according to national guidelines.
* Signed confirmation of participation.

Exclusion Criteria:

* Bilateral breast cancer or suspicion of disseminated cancer
* Unable to understand the information, the planned treatment or follow-up for any reason.
* Earlier radiotherapy towards the thoracic region.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Participant engagement in the decision making process as measured by the Shared Decision Making Questionnaire 9. | Within one week after the consultation
  Minimum value: 0. Maximum value: 100. The higher the value the more patient engagement.

SECONDARY OUTCOMES:
The doctor's perception of patient engagement in the decision making process as measured by the Shared Decision Making Questionnaire doctor 9 | Within one week after the consultation
  Minimum value: 0. Maximum value: 100. The higher the value the more patient engagement.
The participant's fear of cancer recurrence as measured by the Fear of Cancer Recurrence Short form Questionnaire | Within one week after the consultation and again after six months
  Minimum value: 0. Maximum value: 36. The higher the value the more fear of recurrence.
The participant's engagement in the decision making process as measured by the Shared Decision Making Process 4 questionnaire | Within one week after the consultation
  Minimum score: 0. Maximum score: 4. The higher the score the more patient engagement.
The participant's effectiveness in decision making as measured by the Decisional Conflict Scale questionnaire | Before (12 items) and within one week after the consultation (all 16 items)
  Minimum value: 0. Maximum value: 100. The higher the value the more effective decision making.
The participant's regret of the treatment decision as measured by the Decision Regret Scale questionnaire | Six months after the consultation
  Minimum value: 0. Maximum value: 100. The higher the value the more regret.
The participant's engagement in the decision making process as measured by the CollaboRATE questionnaire | Within one week after the consultation
  Minimum score: 0. Maximum score: 9. The higher the value the more patient engagement.
The participant's quality of life as measured by the EORCT QLQ-C30 (version 3.0) questionnaire, only question 29 + 30 | Six months
  Minimum value: 0. Maximum value: 100. The higher the value the more quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Karina D Steffensen, Professor, Study Chair — Vejle Hospital; Stine R Sondergaard, M.D., Principal Investigator — Vejle Hospital
Locations (7):
- Denmark (7):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Herlev
  - Sjaellands University Hospital, Næstved
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No